CLINICAL TRIAL: NCT03236740
Title: Doppler Analysis of Ovarian Stromal Blood Flow Changes After Treatment With Metformin Versus Ethinylestradiol-cyproterone Acetate in Women With Polycystic Ovarian Syndrome
Brief Title: OCP vs Metformin on Ovarian Stromal Blood Flow in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: S.C.B. Medical College and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OG/2017/12
Record Dates: First submitted 2017-07-29; First posted 2017-08-02 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Metformin 500mg bid in morning and evening after meals to be taken for 6 months.
  Interventions: Drug: Metformin Hydrochloride
- OCP (Active Comparator): OCP containing 35 microgram ethinylestradiol and 2-milligram cyproterone acetate to taken from the first day of the menstruation, oral administration of one pill daily for 21 days consecutively, then discontinue using the pill for seven days, and on the eighth day, restart taking the pill. OCP to be taken for 6 months.
  Interventions: Drug: Ethinyl Estradiol-cyprosterone acetate

INTERVENTIONS:
Drug: Ethinyl Estradiol-cyprosterone acetate — Ethinyl Estradiol-cyprosterone acetate in the form of OCPs will be taken cyclically by the participants.
  Arms: OCP
Drug: Metformin Hydrochloride — Metformin Hydrochoride in the form of 500 mg tablets will be taken twice daily by participants.
  Arms: Metformin

SUMMARY:
This study is undertaken to compare the effects of treatment with commonly used OCP containing ethinylestradiol-cyproterone acetate and metformin in women with PCOS. Special attention will be paid to changes in ovarian stromal blood flow by using Color Doppler and they will be correlated with changes in hormonal parameters post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to the Rotterdam criteria

Exclusion Criteria:

* Current or previous use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other hormonal drugs.
* Medical or surgical treatment of PCOS during the previous 3 months
* Presence of other endocrinopathies; except treated hypothyroidism on stable replacement doses of thyroid hormone
* Pregnancy, breastfeeding or desire for pregnancy during study interval (6 months)
* Inability to understand the proposal of the study precluding effective informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in ovarian stromal blood flow by using Doppler | 6 months
  By means of color and power Doppler flow imaging, color signals will be searched in the ovarian stroma away from the ovarian surface and not adjacent to the wall of a follicle. Areas of maximum color intensity, representing the greatest Doppler frequency shifts, will be chosen for pulsed Doppler examination.

SECONDARY OUTCOMES:
Change in BMI as measured in kg/m2 | 6 months
Improvement in hirsutism measured by Modified Ferriman and Gallwey scores | 6 months
Improvement in menstrual cycle pattern | 6 months
Change in waist circumference (cm) | 6 months
Change in blood level of luteinizing hormone [LH] (mIU/ml) and follicle stimulating hormone [FSH] (mIU/ml) | 6 months
Change in blood level of Testosterone (nmol/L) | 6 months
Change in blood level of Sex hormone binding globulin (SHBG) (ng/ml) | 6 months
Change in blood levels of Dehydroepiandrosterone sulfate (DHEAS) level (microgram/dl) | 6 months
Changes in fasting serum insulin levels (mIU/L) | 6 months
Changes in fasting serum glucose levels (mg/dL) | 6 months
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Priyadarshini Tripathy, MD, Principal Investigator — SCB Medical College
Locations (1):
- SCB Medical College, Cuttack, Odisha, India